CLINICAL TRIAL: NCT04178447
Title: An Open-label, Multi-center Trial to Evaluate the Pharmacokinetic Profile of Glepaglutide After a Single Subcutaneous Injection in Subjects With Varying Degrees of Renal Function
Brief Title: Pharmacokinetic Profile of Glepaglutide After a Single Injection in Subjects With Varying Degrees of Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zealand Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ZP1848-18131; 2019-001466-15 (EudraCT Number)
Record Dates: First submitted 2019-11-25; First posted 2019-11-26 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-03

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Intervention Model Description: If only Part A will be conducted total subjects of 16 will be enrolled if Part B also will be conducted up to 48 subjects will be enrolled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1: ESRD subjects not on dialysis or severe RI (Experimental): subjects with eGFR <15 mL/min/1.73 m2) or (eGFR 15 to <30 mL/min/1.73 m2)
  Interventions: Drug: Glepaglutide
- Group 2: normal renal function (Experimental): subjects with eGFR ≥90 mL/min/1.73 m2
  Interventions: Drug: Glepaglutide
- Group 3: moderate RI (Experimental): subjects with eGFR 30 to <60 mL/min/1.73 m2
  Interventions: Drug: Glepaglutide
- Group 4: mild RI (Experimental): subjects with eGFR 60 to <90 mL/min/1.73 m2
  Interventions: Drug: Glepaglutide

INTERVENTIONS:
Drug: Glepaglutide — Single dose of Glepaglutide 10 mg
  Other Names: ZP1848

SUMMARY:
This is two stage design, open-label, multi-center, non-randomized trial evaluating the PK of a single, subcutaneous dose of 10 mg glepaglutide in subjects with varying degrees of renal function. The renal function will be calculated by the estimated glomerular filtration rate (eGFR) according to the Modification of Diet in Renal Disease (MDRD) equation.

ELIGIBILITY:
Inclusion Criteria:

* All subjects

  1. Able to understand and willing to sign the informed consent
  2. eGFR values as defined in in the arms
  3. Willing and able to comply with the study requirements
  4. Male and female subjects age 18 to 70 years (both inclusive) at the time of informed consent
  5. BMI 20.0 - 30.0 kg/m2 both inclusive
  6. Must be willing to comply with the contraception, sperm-donation requirements, and study restrictions.

     Renally Impaired Subjects (in Addition)
  7. Subject has a stable disease, including disease(s) associated with renal impairment, under medical control (ie, no changes in medication within 30 days prior to study drug administration). Stable renal impairment, defined as no clinically significant change in disease status within 3 months before screening.

Exclusion Criteria:

All Subjects

1. Suspicion of hypersensitivity, intolerance, or allergy to glepaglutide
2. History of alcohol or drug abuse
3. Clinically relevant abnormal medical history, abnormal findings on physical examination, vital signs, clinically significant abnormalities on 12-lead ECG, or laboratory tests at Screening that the Investigator judges as likely to interfere with the objectives of the study or the safety of the subject except for conditions associated with renal impairment in subjects with renal impairment
4. Uncontrolled treated/untreated hypertension (defined as a mean of 3 repeated measurements for systolic blood pressure ≥ 180 mmHg and/or diastolic blood pressure ≥ 110 mmHg); current or documented history of repeated clinically significant hypotension or severe episodes of orthostatic hypotension (systolic blood pressure < 90 mmHg and/or diastolic blood pressure < 50 mmHg)
5. Acute illness within 14 days prior to dosing unless mild in severity and approved by the Investigator and Sponsor's medical representative
6. Presence of active infection requiring antibiotics. Ingestion of alcohol within 72 hours prior to study drug administration and during PK sampling period including Follow-Up
7. Participation in another investigational drug study within 30 days prior to study drug administration or exposure to more than three new investigational agents within 12 months prior to study drug administration
8. Previous exposure to GLP-1, GLP-2, human growth hormone, somatostatin, or analogues thereof within 3 months prior to Screening. Use of dipeptidyl peptidase-4 inhibitors within 3 months prior to Screening
9. Previous exposure to glepaglutide
10. Donation or loss of more than 450 mL blood during the 3 months before the start of Screening
11. Female subjects who are breastfeeding, pregnant, or planning to become pregnant during the study
12. Positive serology for hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (anti-HCV) or human immunodeficiency virus antibodies (anti-HIV)-1/2, unless the absence of an active hepatitis B/C infection is confirmed by a polymerase chain reaction (PCR) test, at Screening
13. Positive urine screen of drugs of abuse (if not due to concomitant medication) or alcohol breath test at Screening and/or Day -1
14. Legal incapacity or limited legal capacity

    Renally Impaired Subjects (in Addition)
15. Acute renal failure (as judged by the Investigator)
16. Renal impairment requiring dialysis
17. History of kidney transplant regardless of functionality
18. Serum albumin concentration <25 g/L
19. Haemoglobin concentration <100 g/L
20. Medications known to affect the elimination of serum creatinine (e.g., trimethoprim or cimetidine) and competitors of renal tubular secretion (e.g., probenecid) within 60 days prior to study drug administration

    Subjects With Normal Renal Function (in Addition)
21. Significant medical history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, haematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the Investigator -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2020-07-14 (Actual); Study Completion 2020-07-14 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic Variables | 11 days
  AUC0-168 area under the concentration-time curve (AUC) from time 0 to 168 hours
  Cmax maximum observed plasma concentration

SECONDARY OUTCOMES:
Safety Variables | 11 days
  Number of subject with AE/SAE as a measure of safety and tolerability

CONTACTS AND LOCATIONS:
Locations (3):
- Hungary (2):
  - Fázis I-es Klinikai Farmakológiai, Budapest
  - Szent Imre Egyetemi Oktatókórház, Budapest
- Specjalistyczne Centrum Medyczne - Prywatny Szpital, Krakow, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Agersnap MA, Sonne K, Knudsen KM, Sulowicz W. Pharmacokinetics, Safety, and Tolerability of Glepaglutide, a Long-Acting GLP-2 Analog, in Subjects with Renal Impairment. Clin Pharmacokinet. 2023 Apr;62(4):645-651. doi: 10.1007/s40262-023-01215-9. Epub 2023 Feb 21. PMID 36811175